CLINICAL TRIAL: NCT02933333
Title: G-CSF Alone or Combination With GM-CSF on Prevention and Treatment of Infection in Children With Malignant Tumor: a Prospective, Multicentre, Randomised Controlled Trial
Brief Title: G-CSF Alone or Combination With GM-CSF on Prevention and Treatment of Infection in Children With Malignant Tumor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojun Yuan, chief physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-021
Record Dates: First submitted 2016-10-08; First posted 2016-10-14 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Lymphoma; Neuroblastoma; Hepatoblastoma; Retinoblastoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Neuroblastoma; Hepatoblastoma; Retinoblastoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GM-CSF (Experimental): Eligible patients received subcutaneous GM-CSF 5 μg/kg per day when the first time of absolute neutrophil count [ANC] <1.5*10^9/L after chemotherapy. GM-CSF is given daily for at least 5 days and continued until the ANC reached 1.5*10^9/L for two consecutive days.
  Interventions: Biological: GM-CSF
- G-CSF (Experimental): Eligible patients received subcutaneous G-CSF 5 μg/kg per day when the first time of absolute neutrophil count [ANC] <1.5*10^9/L after chemotherapy. G-CSF is given daily for at least 5 days and continued until the ANC reached 1.5*10^9/L for two consecutive days.
  Interventions: Biological: G-CSF
- G-CSF + GM-CSF (Experimental): Eligible patients received subcutaneous a combination of GM-CSF 5 μg/kg per day and G-CSF 5 μg/kg per day when the first time of absolute neutrophil count [ANC] <1.5*10^9/L after chemotherapy. GM-CSF and G-CSF are given daily for at least 5 days and continued until the ANC reached 1.5*10^9/L for two consecutive days.
  Interventions: Biological: GM-CSF and G-CSF

INTERVENTIONS:
Biological: GM-CSF — Granulocyte-macrophage colony-stimulating factor (GM-CSF) is a hematopoietic CSFs that decrease the duration and severity of neutropenia for patients receiving chemotherapy. GM-CSF is a stimulator of the growth and differentiation of hematopoietic progenitor cells committed to neutrophils, monocytes or eosinophils.
  Arms: GM-CSF
Biological: G-CSF — Granulocyte colony-stimulating factor (G-CSF) is a hematopoietic CSFs that decrease the duration and severity of neutropenia for patients receiving chemotherapy. G-CSF is a relatively specific stimulator of the growth and differentiation of hematopoietic progenitor cells committed to the neutrophil lineage.
  Arms: G-CSF
Biological: GM-CSF and G-CSF — Granulocyte-macrophage colony-stimulating factor (GM-CSF) and granulocyte colony-stimulating factor (G-CSF) are hematopoietic CSFs that decrease the duration and severity of neutropenia for patients receiving chemotherapy. GM-CSF and G-CSF share a number of biologic activities, GM-CSF seems to be more potent against fungi.
  Arms: G-CSF + GM-CSF

SUMMARY:
The purpose of this study is to explore the effect of G-CSF combination with GM-CSF on prevention and treatment of infection in children with malignant tumor.

DETAILED DESCRIPTION:
G-CSF Alone or Combination With GM-CSF on Prevention and Treatment of Infection in Children With Malignant Tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant tumor including acute myeloid leukemia (AML) after complete remission, acute lymphocytic leukemia (ALL) after complete remission, stage III or IV lymphoma after partial remission or complete remission, stage III or IV neuroblastoma (NB) or retinoblastoma (RB).
* Eastern Cooperative Oncology Group performance status ≤ 2.
* Did not receive treatment of CSFs in two weeks.
* Without symptomatic infection and with normal values of C-reactive protein or procalcitonin.
* The first time of ANC < 1.5*10^9/L after chemotherapy.
* More than 24 h after the last chemotherapy.
* The function of liver was normal.

Exclusion Criteria:

* Allergic to GM-CSF or drugs which expressed in Escherichia coli.
* Patients with infection, diabetes or primary immunodeficiency.
* Patients infected with hepatitis B, hepatitis C or HIV.
* Patients confirmed autoimmune thrombocytopenic purpura.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 405 (Estimated)
Dates: Start 2016-09-27 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
assess the incidence of infection in patients after chemotherapy | within 20 days after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Xiaojun, Ph.D, Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Zhai Xiaowen, Ph.D, Principal Investigator — Children's Hospital of Fudan University; Hu Shaoyan, Ph.D, Principal Investigator — Children's Hospital of Soochow University; Fang Yongjun, Ph.D, Principal Investigator — Nanjing Children's Hospital; Wen Hong, Ph.D, Principal Investigator — The First Affiliated of Xiamen University; Wang Hongmei, Ph.D, Principal Investigator — Qianfoshan Hospital; Sun Lirong, Ph.D, Principal Investigator — The Affiliated Hospital of Qingdao University; Li Aimin, Ph.D, Principal Investigator — Yantai Yuhuangding Hospital; Gao Fei, Ph.D, Principal Investigator — Shandong Proincial Hospital; Liu Wei, Ph.D, Principal Investigator — Zhengzhou Children's Hospital; Liang Changda, Master, Principal Investigator — Jiangxi Proincial Children's Hospital; Pan Kaili, Master, Principal Investigator — Northwest Women's Hospital
Locations (7):
- China (7):
  - The First Affiliated of Xiamen University, Xiamen, Fujian
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Shandong Province Qianfoshan Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital affiliated to Shanghai Jiaotong University school of medicine, Shanghai, Shanghai Municipality
  - Northwest Women's Hospital, Xi'an, Shangxi

IPD SHARING:
Plan to Share IPD: No